CLINICAL TRIAL: NCT02832895
Title: Assessment of Frontal Bone Window for Transcranial Doppler Among Acute Brain Injured Patients in Intensive Care Units: a Prospective Study.
Brief Title: Frontal Bone Window in ICUF (FBW-ICU)
Acronym: FBW-ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Conducting an interim analysis that allowed with the number of patients included of 150 to meet the objectives of this research
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9489; 2014-A01436-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Acute Brain Injury
Keywords: Adults; Frontal bone window; Transcranial doppler
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Doppler examination (Experimental): Transcranial Doppler examination
  Interventions: Other: Transcranial doppler examination

INTERVENTIONS:
Other: Transcranial doppler examination — Assessment of frontal bone window for transcranial doppler

SUMMARY:
Transcranial doppler (TCD) is an established tool for monitoring flows in intracranial cerebral arteries. Its use is recommanded in the last guidelines on traumatic brain injury. The temporal bone window (TBW) is limited in evaluating flow in the anterior cerebral arteries (ACA) because of an unfavorable insonation angle. Thereby TCD could be unfit to detect a segmental lesion on the anterior cerebral arteries (ACA).

The frontal bone window (FBW) is a promising approach in evaluating flows in the ACA. However, the utility of the FBW for patients with acute brain injury (ABI) in ICU has not been yet determined.

The goal of the present study is to determine the rate of detection of the ACA by using the FBW in patients with ABI in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Membership in a health insurance scheme
* Patients with an acute cerebral pathology
* Hospitalized patients in a supportive care unit of Montpellier University Hospital
* Be able to benefit from transcranial doppler within 3 days of admission

Exclusion Criteria:

* Clinical suspicion of encephalic death
* Known allergy to ultrasound gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
measures of ACA flow velocities threw the frontal bone window | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Camille CM Maury, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France